CLINICAL TRIAL: NCT00573157
Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Atacicept in Subjects With Lupus Nephritis in Combination With Mycophenolate Mofetil Therapy.
Brief Title: The Efficacy and Safety of Atacicept in Combination With Mycophenolate Mofetil Used to Treat Lupus Nephritis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to unanticipated safety issues
Sponsor: EMD Serono (Industry)
Collaborators: ZymoGenetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28113; 493G01
Record Dates: First submitted 2007-12-11; First posted 2007-12-14 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Lupus Nephritis
Keywords: nephritis; atacicept
MeSH Terms: conditions — Lupus Nephritis; Nephritis | interventions — TACI receptor-IgG Fc fragment fusion protein; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atacicept Plus Mycophenolate mofetil Plus Corticosteroids (Experimental)
  Interventions: Drug: Atacicept; Drug: Mycophenolate mofetil; Drug: Corticosteroids
- Placebo Plus Mycophenolate mofetil Plus Corticosteroids (Placebo Comparator)
  Interventions: Drug: Mycophenolate mofetil; Drug: Placebo; Drug: Corticosteroids

INTERVENTIONS:
Drug: Atacicept — Atacicept will be administered at a dose of 150 milligram (mg) subcutaneously (SC) twice weekly for 4 weeks followed by maintenance dose of 150 mg SC once weekly for 48 weeks.
  Arms: Atacicept Plus Mycophenolate mofetil Plus Corticosteroids
Drug: Mycophenolate mofetil — MMF will be administered orally with a starting dose of 500 mg twice daily for 1 week, will be increased to 1000 mg twice daily for 1 week, then it will be adjusted to 1500 mg or lower twice daily as per investigator's discretion.
Drug: Placebo — Placebo will be administered at a dose of 150 mg SC twice weekly for 4 weeks followed by 150 mg SC once weekly for 48 weeks.
  Arms: Placebo Plus Mycophenolate mofetil Plus Corticosteroids
Drug: Corticosteroids — High dose CS of 0.8 mg per kilogram per day or maximum of 60 mg per day prednisone or prednisone equivalent, whichever is less will be administered for 4 Weeks and will be tapered to 7.5 to 10 mg/day up to Week 12.

SUMMARY:
The purpose of this study is to learn whether atacicept treatment leads to improvement in kidney function in subjects with active lupus nephritis in combination with mycophenolate mofetil (MMF) and corticosteroids. The study was sponsored by Merck Serono International; operational oversight was provided by ZymoGenetics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus (SLE) satisfying at least 4 out of the 11 American College of Rheumatology (ACR) criteria (Appendix B)
* Renal biopsy performed consistent with active International Society of Nephrology/Renal Pathology Society (ISN/PRS) class III or IV lupus nephritis

Exclusion Criteria:

* Estimated glomerular filtration rate (GFR) less than or equal to (<=) 30 milliliter per minute (mL/min) per 1.73 square meter (m^2)
* Active central nervous system SLE deemed to be severe or progressive and/or associated with significant cognitive impairment
* Any treatment with MMF, azathioprine, or cyclophosphamide within the last 6 months, or known hypersensitivity to MMF or atacicept.
* Any prior treatment with abatacept, rituximab, belimumab, or other B cell modulating agents.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (20):
- United States (12):
  - Tulane University Hospital and Clinic Department of Internal Medicine, New Orleans, Louisiana
  - Northwest Louisiana Nephrology Research, Shreveport, Louisiana
  - Wayne State University Lupus Database Departments of Internal Medicine and Obstetrics & Gynecology Division of Rheumatology Wayne State University School of Medicine, Detroit, Michigan
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Seligman Center for Advanced Therapeutics, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rheumatology Clinical Research Unit, Division of Rheumatology University Hospitals Case Medical Center, Beachwood, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Southwest Rheumatology and Research Group, LLC, Middleburg Heights, Ohio
  - 1711 St. Julian Place, Columbia, South Carolina
  - ACME Research, LLC, Orangeburg, South Carolina
- Institute of Rheumatology, Prague, 128 50, Czechia
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Kedah
  - Hospital University Kebangsaan Malaysia, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Pulau Pinang, Pulau Pinang
- Singapore (2):
  - Changi General Hospital, Singapore
  - Singapore General Hospital, Singapore
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Ginzler EM, Wax S, Rajeswaran A, Copt S, Hillson J, Ramos E, Singer NG. Atacicept in combination with MMF and corticosteroids in lupus nephritis: results of a prematurely terminated trial. Arthritis Res Ther. 2012 Feb 7;14(1):R33. doi: 10.1186/ar3738. PMID 22325903

RESULTS

PARTICIPANT FLOW:
Groups:
- Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids: Atacicept was administered subcutaneously (SC) at a loading dose of 150 milligram (mg) twice weekly for 4 weeks followed by maintenance dose of 150 mg SC once weekly for 48 weeks. MMF was administered orally with a starting dose of 500 mg twice daily for 1 week, increased to 1000 mg twice daily for 1 week, then adjusted to 1500 mg or lower twice daily as per investigator's discretion. High dose corticosteroids (CS) of 0.8 mg per kilogram per day or maximum of 60 mg per day prednisone or prednisone equivalent, whichever was less was administered for 4 Weeks and tapered to 7.5 to 10 mg/day up to Week 12.
- Placebo Plus Mycophenolate Mofetil Plus Corticosteroids: Placebo was administered SC at a loading dose of 150 mg twice weekly for 4 weeks followed by maintenance dose of 150 mg SC once weekly for 48 weeks. MMF was administered orally with a starting dose of 500 mg twice daily for 1 week, increased to 1000 mg twice daily for 1 week, then adjusted to 1500 mg or lower twice daily as per investigator's discretion. High dose CS of 0.8 mg per kilogram per day or maximum of 60 mg per day prednisone or prednisone equivalent, whichever was less was administered for 4 Weeks and tapered to 7.5 to 10 mg/day up to Week 12.
Period: Overall Study
Arm/Group | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids
Started | 4 | 2
Completed | 0 | 0
Not Completed | 4 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all the participants randomized in the trial.
Groups:
- Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids: Atacicept was administered SC at a loading dose of 150 mg twice weekly for 4 weeks followed by maintenance dose of 150 mg SC once weekly for 48 weeks. MMF was administered orally with a starting dose of 500 mg twice daily for 1 week, increased to 1000 mg twice daily for 1 week, then adjusted to 1500 mg or lower twice daily as per investigator's discretion. High dose CS of 0.8 mg per kilogram per day or maximum of 60 mg per day prednisone or prednisone equivalent, whichever was less was administered for 4 Weeks and tapered to 7.5 to 10 mg/day up to Week 12.
- Total: Total of all reporting groups
Arm/Group | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.3) | 36.0 (25.5) | 36.5 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Complete Renal Response (CRR), Partial Response, and Non-response
Description: Complete renal response (CRR): from baseline, a return to within 10% of normal for renal function (assessed by calculated glomerular filtration rate [GFR]), improvement in proteinuria (urine protein/creatinine ratio <0.5) & resolution of hematuria. Partial response (PR): from baseline, a <= 10% worsening in renal function ( by calculated GFR); 50% improvement in proteinuria (assessed by urine protein/creatinine ratio) & resolution of hematuria, Non-response (NR): Neither criteria for CR or PR was met. Subjects were also deemed NR if they had treatment failure, regardless of CR or PR status. Subjects cannot be treatment failures. A response of CRR was confirmed if the Week 52 value is CRRand if the Week 48 value is CRR and at least 4 weeks apart from Week 52 /if the Week 48 value was missing/ less than 4 weeks from Week 52, then the Week 56 response must be CRR - if the Week 52 value was missing, then Week 48 and Week 56 must be CRR.
Time Frame: At Week 52
Population: Due to early termination of the study caused by unanticipated safety issues, the outcome measure was not assessed.
Arm/Group | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Normalization of Renal Function
Time Frame: At Week 52
Population: Due to early termination of the study caused by unanticipated safety issues, the outcome measure was not assessed.
Arm/Group | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With New Lupus Flares
Time Frame: At Week 52
Population: Due to early termination of the study caused by unanticipated safety issues, the outcome measure was not assessed.
Arm/Group | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication to 24-Week follow-up after last dose of trial medication.
Description: A Serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Arm/Group | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids
Serious Adverse Events (participants affected / at risk) | 3/4 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids (N=4) | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids (N=2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept Plus Mycophenolate Mofetil Plus Corticosteroids (N=4) | Placebo Plus Mycophenolate Mofetil Plus Corticosteroids (N=2)
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 0
Injection site haematoma (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Blood immunoglobulin G decreased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to unanticipated safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing results, Institution and Principal Investigator (PI) must first provide Sponsor with a copy of proposed publication for review at least 30 days prior to submission. If Institution and PI do not agree to modification, they shall so notify Sponsor and postpone submission for additional 60 days to allow Sponsor to seek legal remedies or file patent applications. There is a need for coordinated approach to any publication of results from sites for any multi-site study.